CLINICAL TRIAL: NCT04218149
Title: Comparison of the Effects of Serratus Plane Block and Erector Spinae Plane Block on Postoperative Analgesia in Patients Undergoing Unilateral Breast Surgery
Brief Title: Serratus Plane Block vs Erector Spinae Plane Block on Postoperative Analgesia in Patients Undergoing Unilateral Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerim Şahin, research assistant, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS01
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Postoperative Pain
Keywords: serratus plane block, erector spinae plane block, postoperative analgesia
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S (Active Comparator): Serratus plane block with 25 ml %0.25 bupivacaine
  Interventions: Drug: Bupivacaine Injection
- Grup E (Active Comparator): Erector spinae plane block with 25 ml %0.25 bupivacaine
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — Block with bupivacaine

SUMMARY:
Interfacial plan blocks are becoming more widely used for postoperative analgesia because of their easier applicability and less risk of complications. In this study, we aimed to compare the effects of serratus plane block (SPB) and erector spinae plane block (ESPB) on postoperative analgesia in patients undergoing unilateral breast surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age: 18 - 65 years
* unilateral breast surgery

Exclusion Criteria:

* Does not approve the study
* Pregnant
* Emergency
* ASA III-IV
* History of local anesthetic allergy
* Infection in the block area
* Coagulation disorder
* Morbid obesity (body mass index> 40 kg / m²)
* Severe organ failure
* Previous neurological deficit
* Psychiatric disease
* History of chronic pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | Postoperative 24 hours
  Visual analog scale (0-10), <4 is adequate analgesia
Postoperative tramadol consumption | Postoperative 24 hours
  Postoperative opiodi consumption with patient controlled analgesia
Rescue analgesic | Postoperative 24 hours
  If VAS score is 4 or more, paracetamol 1 gr is administered

SECONDARY OUTCOMES:
Analgesia time | Procedure
  Time from block performing to first analgesia requirement

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)